CLINICAL TRIAL: NCT07090200
Title: Rehabilitation Intervention for COPD Combined With Cardiovascular and Cerebrovascular Diseases
Acronym: RI-COPD & CCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Subdecanal,Professor and Director of Respiratory and Critical Care Medicine, Chief Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: XHJY-Chronic disease; 2023ZD0509905 (Other Grant/Funding Number: Research on major national science and technology projects)
Record Dates: First submitted 2025-05-04; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Diseases; Cardiovascular Diseases; Cerebrovascular Diseases
Keywords: prevention; treatment strategies; respiratory diseases; cardiovascular diseases; cerebrovascular diseases
MeSH Terms: conditions — Respiratory Tract Diseases; Cardiovascular Diseases; Cerebrovascular Disorders | interventions — Drug Therapy; Population Groups

STUDY DESIGN:
Intervention Model Description: Firstly, to screen out the high-risk population of COPD combined with cardiovascular and cerebrovascular diseases, COPD with cardiovascular and make a diagnosis. Then, participants were randomized (1:1) to either the optimized or routine group via a computer-generated random number table. The Routine Care Group received treatment for three months and follow-up with medications prescribed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 Report. The Pulmonary Rehabilitation Care Group received the Pulmonary rehabilitation exercise and usual care for three months. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function of the two groups of patients one year after the intervention. And finally, to build a trinity model of rehabilitation management of COPD patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD Pulmonary Rehabilitation Care Group (Experimental): The Pulmonary Rehabilitation Care Group received the Pulmonary rehabilitation exercise and usual care for three months. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function one year after the intervention.
  Interventions: Combination Product: Pulmonary Rehabilitation Care Group
- COPD Routine Care and Sham Comparator Group (Sham Comparator): The Routine Care Group received treatment for three months and follow-up with medications prescribed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 Report. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function of the two groups of patients one year after the intervention.
  Interventions: Other: The Routine Care (Non-Pharmacological and Pharmacological Treatments ) Group

INTERVENTIONS:
Combination Product: Pulmonary Rehabilitation Care Group — participants were randomized (1:1) to either the optimized or routine group via a computer-generated random number table. The Routine Care Group received treatment for three months and follow-up with medications prescribed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 Report. The Pulmonary Rehabilitation Care Group received the Pulmonary rehabilitation exercise and usual care for three months. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function of the two groups of patients one year after the intervention.
  Arms: COPD Pulmonary Rehabilitation Care Group
Other: The Routine Care (Non-Pharmacological and Pharmacological Treatments ) Group — participants were randomized (1:1) to either the optimized or routine group via a computer-generated random number table. The Routine Care Group received treatment for three months and follow-up with medications prescribed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 Report. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function one year after the intervention.
  Arms: COPD Routine Care and Sham Comparator Group

SUMMARY:
Firstly, to screen out the high-risk population of COPD combined with cardiovascular and cerebrovascular diseases, COPD with cardiovascular and make a diagnosis. Then, to evaluate the therapeutic effect of Pulmonary rehabilitation exercise and usual care for three months. And finally, to build a trinity model of rehabilitation management of COPD patients. The objective of this project is to establish and promote the application of diagnostic and treatment norms.

DETAILED DESCRIPTION:
Firstly, to screen out the high-risk population of COPD combined with cardiovascular and cerebrovascular diseases, COPD with cardiovascular and make a diagnosis. Then, participants were randomized (1:1) to either the optimized or routine group via a computer-generated random number table. The Routine Care Group received treatment for three months and follow-up with medications prescribed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 Report. The Pulmonary Rehabilitation Care Group received the Pulmonary rehabilitation exercise and usual care for three months. Next, Observe the changes in the improvement of acute exacerbation frequency (times/year/person)，CAT Scoring and St. George's Respiratory Questionnaire (SGRQ), as well as lung ventilation and diffusion function of the two groups of patients one year after the intervention. And finally, to build a trinity model of rehabilitation management of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Committed to adhering to the study protocol and cooperating with the implementation of the entire research process.
2. Aged 18 years or older, regardless of gender.
3. Signed informed consent form.

Exclusion Criteria:

1. Individuals with severe mental illness.
2. Individuals assessed by medical personnel as having a disease that requires immediate hospitalization or a severe, uncontrollable condition that is life-threatening in the short term.
3. Women who are pregnant, breastfeeding, or using inappropriate contraception methods.
4. Individuals who refuse to cooperate with follow-up questionnaires or specimen collection.
5. Patients currently participating in other interventional clinical drug trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of high-risk and diagnosed individuals with COPD | through study completion, an average of 4 year
  We conducted a cross-sectional screening among a total of 50,000 people, and then calculated the proportion of the high-risk and confirmed COPD patients among the total population. We use COPD questionnaire to screen COPD high-risk groups and make a diagnosis of COPD through pulmonary function test.
the improvement of acute exacerbation frequency (times/year/person) | through study completion, an average of 4 year
  Observe the changes in the improvement of acute exacerbation frequency (times/year/person) after intervention

SECONDARY OUTCOMES:
Blood pressure | through study completion, an average of 4 year
  Based on a comprehensive assessment of the patient's blood pressure, blood sugar, blood lipids, etc., the risk of chronic cardiovascular and cerebrovascular diseases was evaluated. All measurements were conducted in accordance with international standards and units （mmHg）
blood lipids | through study completion, an average of 4 year
  The risk of chronic cardiovascular and cerebrovascular diseases was evaluated. based on a comprehensive assessment of the patient's blood pressure, blood sugar, blood lipids, etc.,All measurements were conducted in accordance with international standards and units（mmol/L）.
FBG(fasting blood-glucose) | through study completion, an average of 4 year
  The risk of chronic cardiovascular and cerebrovascular diseases was evaluated. based on a comprehensive assessment of the patient's blood pressure, blood sugar, blood lipids, etc.,All measurements were conducted in accordance with international standards and units（mmol/L）

OTHER OUTCOMES:
Observe the changes of SGRQ | through study completion, an average of 4 year
  Observe the changes in the improvement of acute exacerbation frequency (times/year/person) after intervention.
Observe the changes in CAT Scoring | through study completion, an average of 4 year
  Observe the changes in CAT Scoring after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China